CLINICAL TRIAL: NCT00626041
Title: U-CHAMP: Urban Cardiovascular Health Assessment and Management Program
Acronym: U-CHAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Dr. Charlotte Jones, University of Calgary
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 03 71550000144
Record Dates: First submitted 2008-01-14; First posted 2008-02-29 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Cardiovascular Diseases; Hypertension; Hyperlipidemia; Hyperglycemia
Keywords: Community pharmacies; Primary care networks; Global risk assessment; Blood pressure screening
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): referral to primary care network for management of blood pressure, lipids and diabetes.
  Interventions: Other: participant referral to primary care network physician

INTERVENTIONS:
Other: participant referral to primary care network physician — blood pressure, cholesterol and hemoglobin A1c screening and management

SUMMARY:
High blood pressure, elevated blood glucose and high cholesterol are related to the increased risk of stroke and heart disease. Many studies have shown that this risk can be significantly reduced by lowering blood pressure, blood glucose and cholesterol levels.

Through a collaborative effort between Calgary Safeway pharmacists and Calgary Health Region family physician PCN's, U-CHAMP will deliver a program to assist in the identification and management of people with elevated blood pressure, blood glucose and cholesterol and through this effort, reduce the risk of heart disease and stroke in the urban Calgary population aged 18-85 years.

DETAILED DESCRIPTION:
Hypertension (HBP) has long been correlated with risk of stroke and other adverse cardiovascular outcomes. Randomized controlled trials of blood pressure lowering have demonstrated at least 30% reductions in stroke incidence and improved mortality. Despite being such a readily modifiable risk, HBP remains under diagnosed and under treated. To address this gap, the A-CHAMP (Airdrie Community Hypertension Awareness and Management Program) was successfully piloted in Airdrie, a community of 20,000 north of Calgary, Alberta. Trained volunteers held BP screening sessions for seniors in local pharmacies and referred hypertensive participants to their GP's and trained pharmacists for blood pressure management. Of the 408 screened participants (40% of all Airdrie seniors), 36.5% had uncontrolled HBP. By program end, systolic BP was decreased by 16.8 mm (+/- 14.6. P <.05) and 56.2% of hypertensive participants had reached the 2006 Canadian Hypertension Guideline targets. Airdrie now holds annual blood pressure screenings organized and run by volunteers, demonstrating the sustainability of this approach to population screening and risk factor management in this setting.

In order to fully realize the benefits of cardiovascular risk reduction, U-CHAMP will be expanded to include a more global risk assessment and management protocol including assessments for dyslipidemias and diabetes in an urban setting.

The purpose of this project is:

* To expand the rural scope of A-CHAMP into a larger urban setting (Calgary).
* To include a more global risk assessment (for both coronary artery disease and stroke) and management including: cholesterol (total and HDL cholesterol) and diabetes (capillary HgA1c when appropriate).
* To effect fully sustainable practice change in the management of hypertension, diabetes and dyslipidemias by establishing collaborative partnerships between pharmacists, Calgary Health Region (CHR) physicians (Primary Care Networks: PCN's), the CHR Chronic Disease Management Program (CDM), and selected hypertensive patients.

Components of U-CHAMP are as follows:

* Screening Clinics:

  * Visit 1: The pharmacist determines if the participant has diabetes then performs a BP assessment using a BpTRU device (VSM MedTech, Vancouver, BC). The participant is invited to sign the consent then six BP readings are taken 1 minute apart in the non-dominant arm, and the last five readings averaged. If the average reading is ≥140/90 mmHg (≥130/80 for diabetics), the participant is invited to return to a second BP clinic within the next 2 weeks.
  * Visit 2: BP is taken as above. If the average BP from both visits is ≥140/90 mmHg (≥130/80 mmHg for those with diabetes), The client is invited to participate in the program.
* Intervention:

  * Visit 2 continued: The pharmacist completes the assessment form which includes: age, personal or family history of cardiovascular disease, known diabetes, hypertension or dyslipidemia, lifestyle issues, medication list, medication allergies, adherence history, adverse events experienced and non-prescription medications used including herbs, vitamins, and supplements.
  * Baseline random capillary Total Cholesterol, HDL (Cholestech -LDX ® (Manthomed) and HgA1c (DCA 2000) are obtained and with all the above information, the Framingham global cardiovascular risk score is calculated (for those without known vascular disease and those without diabetes). If the readings are above target (according to the most recent Canadian Guidelines for hypertension, dyslipidemias and diabetes), participants are encouraged to have their full lipid profile and HgA1c done by their family physician and to record the results in a wallet card provided to them. Counseling about global cardiovascular risk, medications (if applicable), lifestyle information, a hypertension education pamphlet (CHEP 2007 public education) and a wallet card are provided.
  * Participants are referred to their primary care physician for further assessment/management. Assessment information with BP, lipid and HgA1c results and any recommendations (according to latest Canadian Guidelines) including the least expensive drug alternatives, are faxed to the participant's primary care physician.
* Follow-up:

  * Participants are asked to return for follow-up several times during the 6 to 12 month program. Participants are encouraged to follow up with their GP's after each pharmacy visit (if appropriate).
  * At each visit the participant's BP is re-checked. Medication counseling, lifestyle and other information is reinforced and the BP handbook is updated. If appropriate, any lipid, diabetes and global cardiovascular risk assessment data is recorded in the participants' wallet card and is reviewed with them. Counseling about the appropriate target levels is provided. Results of the assessment including recommendations and the pharmacist's comments from each visit are faxed to the participant's physician.
* Final Visit:

  * Participants are encouraged to obtain a full lipid profile through their family physician (if appropriate) just prior to their final pharmacy visit (and bring the results to this final visit) so that their Framingham global cardiovascular risk can be recalculated.

The participant's BP, random capillary Total and HDL cholesterol and HgA1c (if appropriate) are measured. Their current medication list is confirmed and adherence information is reviewed and recorded. The final lipid and diabetes lab data (recorded in the BP handbook) is assessed and the global cardiovascular risk score is re-calculated to assess any changes. A copy of the final assessment is faxed to the participant's primary physician. Participants are encouraged to follow up with their GP.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-85 years
* Signed consent

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure between baseline (average of visits one and two) and program end (final visit). | 12 months

SECONDARY OUTCOMES:
Proportion of screened participants identified as being above blood pressure, cholesterol and blood glucose targets at visit two | 12 months
Proportion of participants that achieve published blood pressure (lipid and diabetes when appropriate) targets by program end | 12 months
Proportion of individuals that obtain both a baseline and end of program full lipid panel | 12 months
Change in Framingham Global Cardiovascular Risk score (in those participants that do not have known vascular disease or diabetes and have a recorded baseline and end-of-study full lipid panel). | 12 months
Proportion of individuals that have changes in drug therapy (new medication and/or dosage increase). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Jones, PhD, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Calgary Safeway Pharmacy - Crowfoot Location, Calgary, Alberta
  - Coop Pharmacy - Crowfoot Location, Calgary, Alberta

REFERENCES:
- [Background] McLean DL, McAlister FA, Johnson JA, King KM, Jones CA, Tsuyuki RT. SCRIP-Hypertension program - Improving blood pressure management in patients with diabetes: The design of the SCRIP-HTN study. Canadian Pharmaceutical Journal 139: 1-4, 2006.
- [Background] British Cardiac Society; British Hypertension Society; Diabetes UK; HEART UK; Primary Care Cardiovascular Society; Stroke Association. JBS 2: Joint British Societies' guidelines on prevention of cardiovascular disease in clinical practice. Heart. 2005 Dec;91 Suppl 5(Suppl 5):v1-52. doi: 10.1136/hrt.2005.079988. No abstract available. PMID 16365341
- See also: Related Info — http://www.hypertension.ca
- See also: Related Info — http://www.heartandstroke.ca